CLINICAL TRIAL: NCT01015833
Title: Phase III Randomized Study of Sorafenib Plus Doxorubicin Versus Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Sorafenib Tosylate With or Without Doxorubicin Hydrochloride in Treating Patients With Locally Advanced or Metastatic Liver Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2011-01989; NCI-2011-01989 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000659348; CALGB-80802 (Other: Alliance for Clinical Trials in Oncology); CALGB-80802 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Advanced Adult Hepatocellular Carcinoma; Recurrent Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v7; Stage IIIA Hepatocellular Carcinoma AJCC v7; Stage IIIB Hepatocellular Carcinoma AJCC v7; Stage IIIC Hepatocellular Carcinoma AJCC v7; Stage IV Hepatocellular Carcinoma AJCC v7; Stage IVA Hepatocellular Carcinoma AJCC v7; Stage IVB Hepatocellular Carcinoma AJCC v7; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin; Pharmacogenomic Testing; Sorafenib

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (doxorubicin hydrochloride, sorafenib tosylate) (Experimental): Patients receive doxorubicin hydrochloride IV on day 1 and sorafenib tosylate PO QD or BID on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, patients may continue to receive sorafenib tosylate PO QD or BID in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Drug: Sorafenib Tosylate
- Arm II (sorafenib tosylate) (Experimental): Patients receive sorafenib tosylate PO QD or BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Drug: Sorafenib Tosylate

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Arm I (doxorubicin hydrochloride, sorafenib tosylate)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This randomized phase III trial studies sorafenib tosylate and doxorubicin hydrochloride to see how well they work compared with sorafenib tosylate alone in treating patients with liver cancer that has spread to nearby tissue or lymph nodes or has spread to other places in the body. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving sorafenib tosylate together with doxorubicin hydrochloride is more effective than sorafenib tosylate alone in treating liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the overall survival (OS) of patients treated with sorafenib (sorafenib tosylate) and doxorubicin (doxorubicin hydrochloride) to that of those treated with sorafenib.

SECONDARY OBJECTIVES:

I. Compare time to progression (TTP) of patients treated with sorafenib and doxorubicin to that of those treated with sorafenib.

II. Compare progression-free-survival (PFS) of patients treated with sorafenib and doxorubicin to that of those treated with sorafenib.

III. Compare tumor response using Response Evaluation Criteria in Solid Tumors (RECIST) criteria of patients treated with sorafenib and doxorubicin to that of those treated with sorafenib.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive doxorubicin hydrochloride intravenously (IV) on day 1 and sorafenib tosylate orally (PO) once daily (QD) or twice daily (BID) on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, patients may continue to receive sorafenib tosylate PO QD or BID in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive sorafenib tosylate PO QD or BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically proven hepatocellular carcinoma; known mixed histology (e.g. hepatocellular carcinoma plus cholangiocarcinoma) or fibrolamellar variant is not allowed
* Patients must have locally advanced or metastatic disease; locally advanced disease is defined as disease deemed to be unresectable or non-eligible for transplant without distant metastases
* Lesions must be accurately measurable in at least one dimension (longest diameter to be recorded) as >= 2 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan
* No prior adjuvant sorafenib or other v-RAF-1 murine leukemia viral oncogene homolog (Raf)/vascular endothelial growth factor (VEGF) inhibitors; other prior adjuvant therapy is allowed if completed > 6 months prior to registration with documented recurrence of hepatocellular carcinoma (HCC)
* Patients may have been treated with loco regional therapies provided that they either have:

  * A target lesion that has not been subjected to local therapy or
  * The target lesion(s) within the field of the local therapy has shown an increase of >= 20% in the size since last treatment

    * Such therapy must be completed at least 4 weeks prior to registration; patients that have received palliative radiation therapy to the bone need not wait 4 weeks to begin protocol therapy
* Prior therapies allowed include the following:

  * Bland embolization, radiation, radioactive microspheres, etc
  * Chemoembolization using any chemotherapy (except, see below)
  * Chemoembolization drug-eluting beads using doxorubicin
  * Prior therapy with chemoembolization using doxorubicin in the non drug eluting beads form is NOT allowed
* No prior systemic therapy for metastatic disease
* No prior exposure to systemic doxorubicin administered intravenously
* Antiviral treatment is allowed, however interferon therapy must be stopped at least 4 weeks prior to registration
* Allografts are not allowed: no prior history of any allograft, including but not limited to liver and bone marrow transplants
* Patients must have completed any major surgery >= 4 weeks from registration
* Concomitant treatment with Rifampin or St John's wort is not allowed; patients should discontinue these drugs at least 4 weeks prior to registration
* No known central nervous system (CNS) tumors including brain metastases
* No clinically significant gastrointestinal bleeding events requiring intervention, transfusion, or admission to hospital within 30 days prior to registration
* Patients with a history of hypertension should be well controlled (< 140/90 mmHg) on a regimen of anti-hypertensive therapy
* Significant history of cardiac disease is not allowed:

  * Congestive heart failure > class II New York Heart Association (NYHA)
  * Myocardial infarction within 6 months prior to registration
  * Serious myocardial dysfunction, defined as scintigraphically (multigated acquisition scan [MUGA], myocardial scintigram) determined absolute left ventricular ejection fraction (LVEF) below 45% or an LVEF on echocardiogram (ECHO) below the normal limit at the individual institution
* No history of bleeding diathesis
* Patients receiving combination anti-retroviral therapy for human immunodeficiency virus (HIV) are excluded from the study
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Pregnancy/nursing status: women who are pregnant should not go on study; women should not breastfeed while participating in this study
* Granulocytes >= 1,500/uL
* Hemoglobin >= 8.5 g/dL; patients with recent or ongoing gastrointestinal bleed may not be transfused to reach the entry hemoglobin of 8.5 g/dL; physicians should ensure patients requiring transfusion prior to registration do not have an occult or clinically apparent gastrointestinal bleed
* Platelets >= 75,000/uL
* Creatinine =< 1.5 x upper limit of normal (ULN) (or creatinine clearance calculated >= 60 cc/minute)
* Child-Pugh score A; patients must meet all laboratory value requirements
* Bilirubin =< 3 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 5 x ULN
* Prothrombin time (PT)-international normalized ratio (INR) =< 1.7 (not required for patients on anticoagulation agents; patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2010-02-15 (Actual); Primary Completion 2015-05-21 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan K Abou-Alfa, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (673):
- United States (659):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - East Bay Medical Oncology Hematology Medical Associates Inc-Pleasant Hill, Pleasant Hill, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - University of Colorado Hospital, Aurora, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center -Washington DC, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Advent Health - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - York Hospital, York Village, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Veterans Administration, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Hematology Oncology Associates of Central New York-Liverpool, Liverpool, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Mountain Radiation Oncology PA, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Transylvania Regional Hospital, Brevard, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Mission Hospital McDowell, Marion, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma-Lakeside, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Tech University Health Sciences Center-El Paso, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
- Canada (13):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Fundacion De Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Quintanilha JCF, Geyer S, Etheridge AS, Racioppi A, Hammond K, Crona DJ, Pena CE, Jacobson SB, Marmorino F, Rossini D, Cremolini C, Sanoff HK, Abou-Alfa GK, Innocenti F. KDR genetic predictor of toxicities induced by sorafenib and regorafenib. Pharmacogenomics J. 2022 Dec;22(5-6):251-257. doi: 10.1038/s41397-022-00279-3. Epub 2022 Apr 28. PMID 35484400
- [Derived] Abou-Alfa GK, Shi Q, Knox JJ, Kaubisch A, Niedzwiecki D, Posey J, Tan BR Jr, Kavan P, Goel R, Lammers PE, Bekaii-Saab TS, Tam VC, Rajdev L, Kelley RK, El Dika I, Zemla T, Potaracke RI, Balletti J, El-Khoueiry AB, Harding JJ, Suga JM, Schwartz LH, Goldberg RM, Bertagnolli MM, Meyerhardt J, O'Reilly EM, Venook AP. Assessment of Treatment With Sorafenib Plus Doxorubicin vs Sorafenib Alone in Patients With Advanced Hepatocellular Carcinoma: Phase 3 CALGB 80802 Randomized Clinical Trial. JAMA Oncol. 2019 Nov 1;5(11):1582-1588. doi: 10.1001/jamaoncol.2019.2792. PMID 31486832

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate): Patients receive 60 mg/m2 doxorubicin hydrochloride IV on day 1 and 400 mg sorafenib tosylate PO QD or BID on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses, patients may continue to receive sorafenib tosylate PO QD or BID in the absence of disease progression or unacceptable toxicity.
- Arm II (Sorafenib Tosylate): Patients receive 400 mg sorafenib tosylate PO QD or BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) | Arm II (Sorafenib Tosylate)
Started | 180 | 176
Completed | 167 | 171
Not Completed | 13 | 5
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Symptomatic deterioration | 0 | 1
Not completed — Other | 5 | 1
Not completed — Motor Vehicle Accidents | 1 | 0
Not completed — Did not start treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) | Arm II (Sorafenib Tosylate) | Total
Number analyzed (Participants) | 180 | 176 | 356
Age, Continuous [Median (Full Range); unit: years] | 62 [22 to 81] | 62 [31 to 85] | 62 [22 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 153 | 153 | 306
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 32 | 29 | 61
  United States | 148 | 147 | 295

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death from any cause. The median OS was estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) | Arm II (Sorafenib Tosylate)
Number analyzed (Participants) | 180 | 176
month | 8.9 [7.1 to 10.8] | 10.5 [7.6 to 13.8]
Statistical Analysis 1: Comparison: Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) vs Arm II (Sorafenib Tosylate); Test type: Superiority; p = 0.24, t-test, 1 sided; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.8 to 1.4]

2. Secondary Outcome: Incidence of Toxicities, as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicity is defined as a grade 3 or higher adverse events that is classified as either possibly, probably, or definitely related to study treatment. The assignment of attribution to study treatment and grade (or degree of severity) of the adverse event are classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. The percentage of patients with a maximum grade 3 or higher adverse event at least possibly related to the study treatment are reported below.
Time Frame: Up to 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) | Arm II (Sorafenib Tosylate)
Number analyzed (Participants) | 180 | 176
percentage of patients
  Fatigue | 10 | 7
  Hypertension | 3 | 13
  White blood cells | 11 | 0
  Neutrophils | 33 | 0
  Platelets | 14 | 1
  Hand Foot Syndrome | 10 | 14

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from study entry to earliest date of disease progression. Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: The appearance of one or more new lesions is also considered progression).
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) | Arm II (Sorafenib Tosylate)
Number analyzed (Participants) | 180 | 176
months | 4.0 [3.2 to 5.0] | 3.9 [2.9 to 4.8]
Statistical Analysis 1: Comparison: Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) vs Arm II (Sorafenib Tosylate); Test type: Superiority; p = 0.98, t-test, 1 sided; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.72 to 1.2]

4. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression (TTP) is defined as the time from on study to progression. Progression is defined by the RECIST criteria as Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: The appearance of one or more new lesions is also considered progression). Median and 95% confidence intervals are provided for each arm below.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) | Arm II (Sorafenib Tosylate)
Number analyzed (Participants) | 180 | 176
months | 4.1 [3.25 to 5.00] | 3.8 [2.92 to 4.50]

5. Secondary Outcome: Best Overall Response Rate
Description: Best Overall Response Rate is defined as is the best response recorded from the start of the treatment until disease progression/recurrence. Complete Response: Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: The appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum diameters while on study.
Time Frame: Up to 3 years
Population: Patients who started treatment and had follow-up assessments were included in this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) | Arm II (Sorafenib Tosylate)
Number analyzed (Participants) | 150 | 150
percentage of patients | 7.3 | 3.3

ADVERSE EVENTS:
Time Frame: Up to 3 years.
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who completed the study. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) | Arm II (Sorafenib Tosylate)
All-Cause Mortality (participants affected / at risk) | 12/167 | 16/171
Serious Adverse Events (participants affected / at risk) | 71/167 | 57/171
Other Adverse Events (participants affected / at risk) | 146/167 | 151/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) (N=167) | Arm II (Sorafenib Tosylate) (N=171)
Anemia (Blood and lymphatic system disorders) | 9 (10) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 22 (24) | 28 (33)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (3) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 27 (28) | 13 (15)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4)
Esophagitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 17 (17) | 4 (4)
Nausea (Gastrointestinal disorders) | 34 (36) | 24 (29)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (6)
Death NOS (General disorders) | 4 (4) | 7 (7)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 49 (56) | 32 (38)
Fever (General disorders) | 2 (2) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (2)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bone infection (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3) | 1 (1)
Lung infection (Infections and infestations) | 6 (6) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 2 (2)
Skin infection (Infections and infestations) | 2 (2) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (3) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 6 (6)
Blood bilirubin increased (Investigations) | 8 (9) | 7 (7)
Creatinine increased (Investigations) | 3 (3) | 0 (0)
Ejection fraction decreased (Investigations) | 3 (3) | 1 (1)
Haptoglobin decreased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 2 (2) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (6) | 2 (3)
Neutrophil count decreased (Investigations) | 31 (32) | 0 (0)
Platelet count decreased (Investigations) | 35 (38) | 20 (24)
Weight loss (Investigations) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 10 (10) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 14 (14) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 10 (10) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 (16) | 10 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 21 (25) | 16 (17)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Doxorubicin Hydrochloride, Sorafenib Tosylate) (N=167) | Arm II (Sorafenib Tosylate) (N=171)
Anemia (Blood and lymphatic system disorders) | 10 (11) | 8 (8)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (7) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (5) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 2 (3)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 7 (7) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (4)
Hypothyroidism (Endocrine disorders) | 5 (14) | 4 (18)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 59 (156) | 75 (205)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (3) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (6)
Dental caries (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 68 (203) | 73 (256)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 54 (126) | 31 (45)
Nausea (Gastrointestinal disorders) | 59 (167) | 64 (179)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (5)
Chills (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 4 (6) | 2 (2)
Fatigue (General disorders) | 111 (427) | 104 (407)
Fever (General disorders) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (5) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cecal infection (Infections and infestations) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (2) | 1 (1)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (7) | 6 (10)
Alkaline phosphatase increased (Investigations) | 5 (6) | 9 (13)
Aspartate aminotransferase increased (Investigations) | 12 (15) | 15 (25)
Blood bilirubin increased (Investigations) | 9 (10) | 10 (14)
CD4 lymphocytes decreased (Investigations) | 1 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Ejection fraction decreased (Investigations) | 14 (29) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 3 (4) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (15) | 9 (20)
Neutrophil count decreased (Investigations) | 58 (110) | 11 (69)
Platelet count decreased (Investigations) | 67 (199) | 62 (348)
Weight loss (Investigations) | 1 (1) | 4 (6)
White blood cell decreased (Investigations) | 11 (13) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (8) | 11 (16)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (12) | 9 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (7) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 7 (13) | 11 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (15) | 11 (16)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (3)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (10) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 12 (16)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 57 (197) | 68 (215)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 8 (16) | 7 (9)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 49 (172) | 68 (316)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (15) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less